CLINICAL TRIAL: NCT02608749
Title: Osteoporosis and Fall Prevention High Risk Population Intervention and Follow up in the Metropolitan Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201402022RINB
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Osteoporosis; Fracture
Keywords: Osteoporosis; Fall; Fracture; Sacopenia; Body Composition
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Delivery of Health Care, Integrated; Home Care Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IC (Experimental): Integrated care (IC)
  Interventions: Behavioral: Integrated care (IC)
- LEE (Experimental): Lower extremity exercise (LEE)
  Interventions: Behavioral: Lower extremity exercise (LEE)
- HC (Experimental): Home care (HC)
  Interventions: Behavioral: Home care (HC)

INTERVENTIONS:
Behavioral: Integrated care (IC) — Integraded care (IC) Weekly professional led exercise program for 90 mins with reinforcemen on osteoporosis related educations and caremangements from study educational booklet and CD rom for 3-month. The exercise program included 15 minutes warm up with 10 minute brisk walks followed by gentle stretching. Resistance training (20-30 minutes) was provided with rubber band and bottled water (0.6-1L) as weight for major muscles of upper and lower limbs. Balance training were also provided for 10 minutes with tandem gaits and one leg standing, step up and down stairs, toe walking and heel walking.
  Arms: IC
Behavioral: Lower extremity exercise (LEE) — Lower extremity exercise (LEE) group subjects were invited to BB site to receive 2 sessions of 45-mintute training using isotonic strength training machines on major muslce groups each week. The intensity is set at 60-80% of 1 repetition maximum (RM). Evaluation of the exercise protocol are repeated every 2 weeks for individualized adjustments by trained physical therapist.
  Arms: LEE
Behavioral: Home care (HC) — Home care (HC) group subjects were invited to LK site. For examining whether the exercise video could help elderly people to maintain their exercise and improve their muscle strength or not, the investigators provided exercise video to subjects, and encouraged them to play this exercise at least 2 hours for one week.
  Arms: HC

SUMMARY:
BACKGROUND: The deterioration of musculoskeletal system imposes significant impact on physical activity in older adults.

METHODS: This was a randomized, parallel-group, prospective study. All participants received education program including home-based exercise. The IC group consisted of different modalities of exercise while the LEE group performed machine-based exercise. Body composition, muscle strength, and physical performance were measured at their baseline and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. older than 50 years of age
2. high risk as defined from one of the following criteria

   * score>=1 on one minute osteoporosis risk questionnaire
   * 10 year predicted fracture risk >=20% for major osteoporosis fracture or >=3% for hip fracture from FRAX
   * fall>=2 times in pass 1 year
3. having a bone mineral density test within one year period
4. having the capability to understand the study and complete the study interventions
5. willing to participate for the intervention and study follow ups

Exclusion Criteria:

1. If patients were unable to meet at least the above inclusion criteria.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Lower extremity extensor power measured by isokinetic resistance equipment | 12 weeks
  Lower extremity extensor power is measured by isokinetic resistance equipment by a trained research assistant with standardized protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan